CLINICAL TRIAL: NCT02652403
Title: Quality of Life, Patient Satisfaction, Quality of Dentures, Masticatory Efficiency, Presence of Temporomandibular Dysfunction and Costs Analysis of Simplified and Conventional Techniques for Complete Denture Fabrication
Brief Title: Simplified Versus Conventional Technique for Complete Denture Fabrication.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Ana Luísa de Barros Pascoal, Principal Investigator, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Simplified versus conventional
Record Dates: First submitted 2016-01-04; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Edentulous
Keywords: Denture, Complete; Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complete conventional dentures (Active Comparator): Complete dentures fabricated by conventional technique.
  Interventions: Device: Complete conventional dentures
- Complete simplified dentures (Active Comparator): Complete dentures fabricated by simplified technique
  Interventions: Device: Complete simplified dentures

INTERVENTIONS:
Device: Complete conventional dentures — The typical operations of conventional technique will be carried out dentures fabrication and clinical appointments and laboratory steps will be necessary until denture insertion:
  Preliminary impression using irreversible hydrocolloid in a stock trays; Individual acrylic resin trays fabrication; Functional impressions using Zinc oxide-eugenol paste and low fusion compound in a individual acrylic resin trays; Maxillary occlusion rims fabrication; Maxillary occlusion rims fabrication adjustments, Centric relation records and transference of the maxillary occlusion rims positions to semiadjustable articulators using a facebow; Setting of teeth in wax; Complete denture wax try-in; Insertion, instructions and postinsertion appointments.
  Other Names: Complete traditional dentures
  Arms: Complete conventional dentures
Device: Complete simplified dentures — For a complete simplified denture fabrication, individual acrylic resin trays fabrication and functional impressions steps will be deleted, and the facebow for transference of the maxillary occlusion rims positions to semiadjustable articulators will be replaced by the table Camper.
  Arms: Complete simplified dentures

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a simplified technique of conventional dentures fabrication, comparing it to a traditional technique, by evaluating the impact of oral health on quality of life, satisfaction of individuals and chewing efficiency as well assessing the quality of prosthetics and TMD. Furthermore, the cost involved in the manufacture of dentures through technique simplified will be compared to the cost involved in the traditional technique.

DETAILED DESCRIPTION:
The traditional technique will be conducted through a protocol used by most dental schools in Brazil and described in some clinical trials as a conventional technique for dentures fabrication. On simplified technical functional molding step is deleted, and thus the orientation planes are made directly on the resulting models of the initial molding alginate, and the mounting of the models is performed in semiadjustable articulators random with the aid of an auxiliary table 15 degrees with semiadjustable articulators fixed to the slope. To evaluate the impact on oral health quality of life of individuals will be used the Brazilian version of Oral Health Impact Profile for edentulous patients (OHIP-Edent) for evaluation of patient satisfaction will use a specific questionnaire assessing the quality of the prostheses will be carried out through a specific exam, to assess the presence of TMD, all subjects will be evaluated through the RDC / TMD, for assessing the efficiency masticatory chewing capsules are used, the costs involved in the manufacture of prostheses will be calculated according to the material consumption used during the making of the prosthesis. All subjects will be assessed before making the prostheses and 90 days after installation of new dentures during this period will be held regular control visits. The data will be evaluated in order descriptive by numbers and proportions, moreover, it will be statistically evaluated by means of suitable tests.

ELIGIBILITY:
Inclusion Criteria:

Edentulous individuals for more than one year and total bimaxillary prosthesis users that need a couple of new prostheses.

Exclusion Criteria:

Pathological changes of alveolar ridges, motor problems and systemic diseases that may influence on the individual's adaptation to the prosthesis.

Ages: 35 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Quality of life | Baseline = day 0
  To assess the impact of oral health on quality of life individuals will be used the Brazilian version of Oral Health Impact Profile for edentulous patients (OHIP-Edent). The inventory shall be applied by a masked examiner.
Patient satisfaction | Baseline = day 0
  Patient satisfaction about complete dentures will be access using a questionnaire that assesses aspects related to overall quality of prosthesis, as well as comfort, aesthetics, retention, phonetics and mastication.
Masticatory efficiency | Three months
  The evaluation of the masticatory efficiency will be conducted through chewing capsules.
Quality of life | Three months
  To assess the impact of oral health on quality of life individuals will be used the Brazilian version of Oral Health Impact Profile for edentulous patients (OHIP-Edent). The inventory shall be applied by a masked examiner.
Patient satisfaction | Three month
  Patient satisfaction about complete dentures will be access using a questionnaire that assesses aspects related to overall quality of prosthesis, as well as comfort, aesthetics, retention, phonetics and mastication.

SECONDARY OUTCOMES:
Costs analysis | Baseline = day 0
  Assessment of the costs involved in the dentures fabrication will be calculated according to the methodology applied by Takanashi et al. 2004.
Quality of dentures | Three months
  Assessment of the technical quality of dentures will be done using an examination that analyzes 14 variables: Selection of artificial teeth; Arrangement of the anterior teeth; Interocclusal distance; Stability of the upper and lower prosthesis; Language space; Centric occlusion; Occlusion during the excursive movements; Retention of upper and lower dentures; Edge of the upper prosthesis extension; Edge of the lower prosthesis extension; facets; Positioning of the posterior teeth.
Temporomandibular dysfunction | Baseline = day 0
  To evaluate the presence of TMD, all subjects will be assessed through RDC / TMD translated and validated to Portuguese by a masked examiner.
Temporomandibular dysfunction | Three month
  To evaluate the presence of TMD, all subjects will be assessed through RDC / TMD translated and validated to Portuguese by a masked examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia dos Santos Calderon, Doctor, Study Director — Universidade Federal do Rio Grande do Norte

REFERENCES:
- [Background] Takanashi Y, Penrod JR, Lund JP, Feine JS. A cost comparison of mandibular two-implant overdenture and conventional denture treatment. Int J Prosthodont. 2004 Mar-Apr;17(2):181-6. PMID 15119869